CLINICAL TRIAL: NCT02904460
Title: Assessment of the Reducting Effect of Dexmedetomidine on the Morphine Use for Severe Burned Patients
Brief Title: Dexmedetomidine for Morphine Consumption Reduction (DEXDOR)
Acronym: DEXDOR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-03Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Burning
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The new progresses relative to sedation-analgesia for resuscitation unit lead to perform a light and cooperative sedation as soon as possible in order to decrease the period of mechanical ventilation. Dexmedetomidine (DEX), which is a central alpha-2 agonist, is the referential hypnotic in this case with a reduction of the morphine-type use.

DEX was mainly studied in the bandage procedures for the burned adult. The aim of this study is to evaluate the reducing effect of DEX on the morphine use in case of severe burnings for adults, to describe the receivers of DEX and to report the procedure of this new molecule.

DETAILED DESCRIPTION:
The new progresses relative to sedation-analgesia for resuscitation unit lead to perform a light and cooperative sedation as soon as possible in order to decrease the period of mechanical ventilation. Dexmedetomidine (DEX), which is a central alpha-2 agonist, is the referential hypnotic in this case with a reduction of the morphine-type use.

DEX was mainly studied in the bandage procedures for the burned adult. The aim of this study is to evaluate the reducing effect of DEX on the morphine use in case of severe burnings for adults, to describe the receivers of DEX and to report the procedure of this new molecule.

This study would manage to develop a protocol using dexmedetomidine to reduce the use of morphine for the sedation-analgesia. It expects a sensitization of physicians about the need to form the nurse crew for the autonomous use of a protocol before performing a new evaluation of sedation-analgesia.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Hospitalised for severe burning (total burned skin surface higher than 20% and/or smoke inhalation and/or severe comorbidities)
* Having received a continued dexmedetomidine administration of at least 24 hours for the case group and having received no dexmedetomidine administration for the control group

Exclusion Criteria:

* Inability to communicate (language barrier, major cognitive disorders)
* Medical contraindication for dexmedetomidine (hepatocellular insufficiency, hypersensibility, grade II or III atrio-ventricular blocks without device, acute brain vascular pathology).
* For the control group, pregnancy is a non-inclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe burned patients cared by the Severe Burned Center between 1st January 2014 and 31 August 2015
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Global consumption of opioids (including per anesthesia for bandage or surgery) during the patient care period, expressed as intravenous morphine per day equivalent, indexed on the weight (mg.kg-1.j-1). | day 20
  mg.kg-1.j-1

SECONDARY OUTCOMES:
Tolerance for dexmedetomidine by hemodynamic | day 20
  mm Hg
Efficiency of analgesia | day 20
  RASS scale

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Reine LOSSER, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France